CLINICAL TRIAL: NCT05541315
Title: A Double-blind, Randomized, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-88260237 in Healthy Participants
Brief Title: A Single Ascending Dose Study of JNJ-88260237 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR109227; 88260237CKD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-09-14; First posted 2022-09-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-88260237 (Experimental): Participants will be randomized into 6 cohorts to receive single oral dose of JNJ-88260237 on Day 1. The doses in each cohort (Cohorts 2 to 4 and 6) will be escalated based on the safety and pharmacokinetics (PK) data of the previous cohort. For Cohort 5, participants will receive a single-dose of JNJ-82260237 in fasted conditions and a single dose of JNJ-82260237 in fed conditions with dosing sequence determined by randomization.
  Interventions: Drug: JNJ-88260237
- Placebo (Placebo Comparator): Participants in Cohorts 1 to 4 and 6 will receive single oral dose of matching placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-88260237 — JNJ-88260237 will be administered orally.
  Arms: JNJ-88260237
Drug: Placebo — Matching placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of a single oral dose of JNJ-88260237 in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Otherwise, healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead electrocardiogram (ECG) evaluations performed at screening
* Body mass index (BMI) within the range 18 to 30 kilogram/meter^2 (kg/m^2) (inclusive)
* A female must be a) not of childbearing potential defined as postmenopausal or permanently sterile
* A female must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 30 days after administration of study intervention
* A male participant must agree not to donate sperm for the purpose of reproduction or plan to father a child during the study and for a minimum of 90 days after receiving study intervention

Exclusion Criteria:

* History of liver (with the exception of Gilbert's syndrome or asymptomatic gallstones) or renal insufficiency (estimated glomerular filtration rate [eGFR] below 90 mL/minute at screening only); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Any history of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin)
* Had major surgery (example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has any surgery planned during the time the participant is expected to participate in the study or within 4 weeks after study intervention administration
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study intervention(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Any current active infections, including localized infections, or any recent history (within 4 weeks prior to administration of study intervention) of active infections, or a history of recurrent, severe, or chronic infections, or otherwise increased risk of infection

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Cohort 1 to 4 and Cohort 6: Number of Participants with Adverse Events (AEs) | Up to Day 14
  Number of participants with AEs will be reported.
Cohort 5: Number of Participants with Adverse Events (AEs) | Up to Day 24
  Number of participants with AEs will be reported.
Cohort 1 to 4 and Cohort 6: Number of Participants with Abnormalities in Vital Signs | Up to Day 7
  Number of participants with abnormalities in vital signs (including body temperature, pulse rate, respiratory rate, and blood pressure) will be reported.
Cohort 5: Number of Participants with Abnormalities in Vital Signs | Up to Day 21
  Number of participants with abnormalities in vital signs (including body temperature, pulse rate, respiratory rate, and blood pressure) will be reported.
Cohort 1 to 4 and Cohort 6: Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Day 7
  Number of participants with abnormalities in ECGs (digital 12-lead ECGs/Holter ECGs) will be reported.
Cohort 5: Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Day 21
  Number of participants with abnormalities in ECGs (digital 12-lead ECGs/Holter ECGs) will be reported.
Cohort 1 to 4 and Cohort 6: Number of Participants with Abnormalities in Clinical Safety Laboratory Parameters | Up to Day 7
  Number of participants with Abnormalities in clinical safety laboratory parameters (including hematology, clinical chemistry, and urinalysis) will be reported.
Cohort 5: Number of Participants with Abnormalities in Clinical Safety Laboratory Parameters | Up to Day 21
  Number of participants with Abnormalities in clinical safety laboratory parameters (including hematology, clinical chemistry, and urinalysis) will be reported.
Cohort 1 to 4 and Cohort 6: Number of Participants with Abnormalities in Physical Examinations | Up to Day 7
  Number of participants with abnormalities in physical examinations will be reported.
Cohort 5: Number of Participants with Abnormalities in Physical Examinations | Up to Day 21
  Number of participants with abnormalities in physical examinations will be reported.

SECONDARY OUTCOMES:
Maximum Observed Whole Blood Concentration (Cmax) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  Cmax is defined as the maximum whole blood concentration of JNJ-88260237.
Time to Reach the Maximum Whole Blood Concentration (Tmax) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  Tmax is defined as the time to reach the maximum whole blood concentration of JNJ-88260237.
Area Under the Whole Blood Concentration Versus Time Curve from Time Zero to Time of the Last Measurable Concentration (AUC [0-Last]) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  AUC (0-Last) is defined as the area under the whole blood concentration versus time curve from time zero to time of the last measurable concentration of JNJ-88260237.
Area Under the Whole Blood Concentration Versus Time Curve from Time Zero to Infinite Time (AUC [0-Infinity]) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  AUC (0-infinity) is defined as the area under the whole blood concentration versus time curve from time zero to infinite time of JNJ-88260237.
Terminal Half-life (T1/2) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  T1/2 is defined as the terminal half-life of JNJ-88260237.
Apparent Oral Whole Blood Clearance (CL/F) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  CL/F is defined as apparent oral whole blood clearance of JNJ-88260237.
Apparent Volume of Distribution (Vz/F) of JNJ-88260237 | Cohort 1 to 4 and Cohort 6: Up to Day 7; Cohort 5: Up to day 21
  Vz/F is defined as the apparent volume of distribution of JNJ-88260237.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency